CLINICAL TRIAL: NCT05793996
Title: Study of the Prevalence of Iron Deficiency Among Hospitalized Patients With HFpEF and the Impact of Ferinject® on Indicators of Quality of Life, Functional Status in Patients With Iron Deficiency
Brief Title: The Prevalence of Iron Deficiency and the Effectiveness of Ferinject® in Patients With HFpEF (ID-HFpEF)
Acronym: ID-HFpEF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-HFpEF
Record Dates: First submitted 2023-03-01; First posted 2023-03-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Heart Failure; Iron Deficiency, Latent
Keywords: HFpEF; iron deficiency; ferric carboxymaltose; Ferinject
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric carboxymaltose; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: 1 (Active Comparator): Drug: Ferinject ® (Ferric carboxymaltose)
  Interventions: Drug: Ferinject
- Comparison Group: 2 (Other): Diet therapy, without drug therapy
  Interventions: Other: Diet therapy
- Control Group: 3 (No Intervention): Without therapy

INTERVENTIONS:
Drug: Ferinject — The calculation of the dose of iron carboxymaltosate (Ferinject ® preparation) for the purpose of correction of iron will be carried out on the basis of the following step-by-step approach: determination of individual iron needs, calculation and administration of iron dose, assessment of the saturation of the patient's body with iron 6 weeks after infusion.
  Other Names: Ferric carboxymaltose
  Arms: Experimental: 1
Other: Diet therapy — Patients will receive diet therapy to correct latent iron deficiency
  Arms: Comparison Group: 2

SUMMARY:
Observational cohort randomized controlled study to study the influence of correction of ID by intravenous injection of ferric carboxymaltose (Ferinject®) on quality of life indicators, functional status in a cohort of patients with HFpEF.

DETAILED DESCRIPTION:
The prevalence of HFpEF among patients admitted to cardiology hospitals will be studied. The study will include patients with NYHA II-III who have signed an informed consent that meets the inclusion/exclusion criteria. The effectiveness of intravenous administration of iron carboxymaltose (Ferinject ® ) to correct iron deficiency and improve the clinical course of HFpEF will be evaluated. A group without iron deficiency will be recruited as a control group (n=30).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study;
* In New York Heart Association (NYHA) II-III functional class due to stable symptomatic chronic heart failure (CHF);
* Left ventricular ejection fraction (LVEF) ≥50%; objective signs of structural and/or functional disorders of the heart consistent with the presence of LV diastolic dysfunction/increased LV filling pressure, including elevated levels of natriuretic peptide;
* Screening ferritin below 100 µg/L, or below 300 µg/L when transferrin saturation (TSAT) is below 20%;
* Screening haemoglobin (Hb) at the time of switching on ( 90-150 g/l).

Exclusion Criteria:

* Uncontrolled arterial hypertension;
* Аnemia not related to iron deficiency;
* Аnemia with a hemoglobin level of less than 90 g/l;
* Less than 1 year after acute myocardial infarction;
* Less than 1 year after acute cerebral circulation disorder;
* Less than 1 year after surgical interventions, including non-cardiac operations and myocardial revascularization (coronary bypass surgery, coronary artery stenting), operations for valvular pathology;
* Chronic alcoholism (including alcoholic heart disease), mental disorders;
* Severe hepatic (increased transaminase levels above the upper three limits of normal) and renal insufficiency (glomerular filtration rate less than 15 ml/min/1.73 m2);
* Known active infection, clinically significant bleeding, active malignancy;
* Severe autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, etc.);
* Severe bronchial asthma, COPD in the acute stage;
* Allergic reactions to medications in the anamnesis, eczema, atopic allergic reaction;
* Blood transfusions and taking erythropoiesis-stimulating drugs during the previous three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome (Combined) | 12 months
  Change of 5 or more points on the Kansas City Cardiomyopathy Questionnaire (KCCQ) (0-100 points)+change in test distance with a 6-minute walk (6MWD - 150 meters or more) by 35 meters or more.
  An increase in the number of points by 5 on the Kansas City Cardiomyopathy Questionnaire scale, increasing the distance on the 6-minute walk test by 35 meters means a better result.
  The absence of changes/decrease in the number of points on the Kansas City Cardiomyopathy Questionnaire scale, the absence of changes/decrease in the distance in the 6-minute walking test means the worst result.

SECONDARY OUTCOMES:
Changing by 5 or more points on the Kansas City Cardiomyopathy Questionnaire (KCCQ 0-100 points) | 6 months
  Change of 5 or more points in the Kansas City Cardiomyopathy Questionnaire (KCCQ) (0-100 points).
  An increase in the number of points by 5 on the Kansas City Cardiomyopathy Questionnaire scale means a better result.
  The absence of changes/decrease in the number of points on the Kansas City Cardiomyopathy Questionnaire scale means the worst result.
Changing in test distance with a 6-minute walk (6MWD 300 meters or more) of 35 meters | 6 months
  Change in the distance when testing a 6-minute walk by 35 meters or more. An increase the distance on the 6-minute walk test by 35 meters or more means a better result.
  The absence of changes/decrease in the distance in the 6-minute walking test means the worst result.
Changing functional class of chronic heart failure (CHF) by New York Heart Association (NYHA I-IV functional classes) | 6 months
  Reduction of the functional class of CHF according to New York Heart Association by 1point means a better result.
  No changes or an increase in the functional class means a worse result.
Hospitalization for heart failure and death from all causes | 12 months
  The absence of hospitalizations for heart failure and death from all causes means a better result. Hospitalization and death from all causes means the worst result.
Changing by 5 or more points according to the Minnesota Heart Failure Quality of Life Questionnaire (MHFLQ) (0-105 points). | 6 months
  A decrease of 5 or more points on the Minnesota Heart Failure Quality of Life Questionnaire (MHFLQ) means a better result.
  The absence of changes/increase in the number of points on the Minnesota Heart Failure Quality of Life Questionnaire (MHFLQ) means the worst result.

CONTACTS AND LOCATIONS:
Overall Officials: Alla A. Garganeeva, M.D., Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No